CLINICAL TRIAL: NCT05252546
Title: A Single-centre, Open, Single-dose, Fixed-sequence Study to Investigate the Effect of Montmorillonite Power or Loperamide on the Pharmacokinetics of Pyrotinib in Healthy Chinese Adult Subjects
Brief Title: Effect of Montmorillonite Power or Loperamide on the Pharmacokinetics of Pyrotinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-DDI-07
Record Dates: First submitted 2022-02-16; First posted 2022-02-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: HER2-positive Recurrent / Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Loperamide

STUDY DESIGN:
Intervention Model Description: Pyrotinib alone and then combined with Montmorillonite Power or Loperamide
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib alone, then pyrotinib + Montmorillonite Power or Loperamide (Experimental): Sequential treatments of pyrotinib alone followed by pyrotinib + Montmorillonite Power or Loperamide, with a washout period in between.
  Interventions: Drug: pyrotinib tablet; Drug: Montmorillonite Power; Drug: Loperamide

INTERVENTIONS:
Drug: pyrotinib tablet — single oral dose of pyrotinib or co-administered with Montmorillonite Power or Loperamide
Drug: Montmorillonite Power — 3 g or one pouch of montmorillonite power 2 hours after pyrotinib administration
Drug: Loperamide — 4 mg of loperamide with pyrotinib followed by 2mg every 2 hours for 2 times for a total of 8mg/day

SUMMARY:
The study will assess the effect of anti-diarrhea drug Montmorillonite Power or Loperamide on the single dose pharmacokinetic parameters of pyrotinib in healthy Chinese subjects. The safety of pyrotinib alone and when co-administered with each drug will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions.
2. Able to complete the study as required by the protocol.
3. Healthy male and female subjects aged 18 to 45 years on the day of signing the informed consent form; appropriate proportion of subjects of different genders (no less than 3 of single gender) required in both groups A and B.
4. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg/m2.
5. Subjects of childbearing potential and their partners have no birth plan and voluntarily take effective contraception during the course of clinical trial until 3 months after the last dose (Female subjects are also required to use highly effective non-drug contraception starting two weeks before study entry and can use contraceptives after study completion).

Exclusion Criteria:

1. Blood donation no less than 400 mL or have blood transfusion within 3 months of dosing.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound or known allergy to pyrotinib, montmorillonite power, loperamide or the excipients;
3. History of drug abuse in the past 5 years, or positive for drug abuse screening;
4. History of alcoholism with alcohol consumption over 14 units per week; heavy smoker; and can't abstain from smoking and alcohol during the study
5. QTcF >470 msec for females or >450 msec for males by 12 lead electrocardiograph;
6. Left ventricular ejection fraction (LVEF) <50% by echocardiography
7. Significant history or clinical manifestation of any neurological, cardiovascular, renal, gastrointestinal, pulmonary, respiratory, metabolic and musculoskeletal disorder, as determined by the Investigator (or designee).
8. Any surgery within 6 months before screening;
9. Intake of hepatotoxic drugs for a long time within 6 months before screening;
10. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months;
11. Subjects who took any drugs that change liver enzymes activity within 28 days before dosing;
12. Subjects who took any prescription drugs, over-the-counter drugs or vitamins, health products or herbal medicine within 14 days before dosing;
13. Clinically significant abnormalities as determined by the Investigator (or designee) in general physical examination, vital signs, laboratory tests, etc.
14. Pregnant or lactating females
15. Positive serology test results for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or human immunodeficiency virus antibody.
16. Subjects who took any beverage or food containing grapefruit, xanthine, caffeine, or alcohol within 48 hours before dosing; strenuous exercise; or other factors which affect drug absorption, distribution, metabolism, excretion, etc
17. Subjects who need to avoid inhibiting intestinal peristalsis, such as patients with flatulence or constipation, or gastrointestinal symptoms such as diarrhea, dry mouth, abdominal distension, anorexia, gastrointestinal spasm, nausea, vomiting, as well as dizziness, headache and fatigue;
18. Those who have special requirements for diet and cannot comply with the diet and corresponding requirements provided by the trial;
19. Those who cannot tolerate venipuncture or with a history of needle-sickness and blood-sickness.
20. Those who have received a live vaccine 2 weeks prior to dosing or are scheduled to be vaccinated within 7 days after study completion.
21. Subjects who, in the opinion of the Investigator should not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Cmax of pyrotinib | Day 1 and Day 9
  Maximum concentration (Cmax) of pyrotinib
AUC of pyrotinib | Day 1 and Day 9
  Area under the plasma concentration versus time curve of pyrotinib

SECONDARY OUTCOMES:
PK parameters （Tmax） of pyrotinib | Day 1 and Day 9
AEs and SAEs | From the first drug administration to 7 days after the last drug administration
  Adverse events and serious adverse events
PK parameters （CL/F） of pyrotinib | Day 1 and Day 9
PK parameters （Vz/F） of pyrotinib | Day 1 and Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang Y, Li D, Zhang T, Xu S, Zhang Y, Zhao K, Li S, Shen K, Li X, Xu P. Evaluation of the pharmacokinetic interactions of montmorillonite powder or loperamide on pyrotinib in healthy volunteers. Front Pharmacol. 2025 May 12;16:1563556. doi: 10.3389/fphar.2025.1563556. eCollection 2025. PMID 40433999